CLINICAL TRIAL: NCT05275192
Title: Utilization of a Videoscope to Improve Clinical Outcomes of Periodontal Regeneration. A Pilot Study
Brief Title: Utilization of a Videoscope in Periodontal Regeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Salvador Nares, DDS, MS, PHD, MBA, Professor and Department Head, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-1311
Record Dates: First submitted 2022-02-04; First posted 2022-03-11 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Chronic Periodontitis
Keywords: Periodontitis; Minimally invasive surgery; Videoscope; Guided tissue regeneration; Stage III, Grade B periodontitis
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Videoscope-assisted periodontal regeneration minimally invasive surgery (Experimental): Videoscope-assisted periodontal regeneration minimally invasive surgery - Test group
  Interventions: Device: Videoscope-assisted periodontal regeneration minimally invasive surgery
- Periodontal regeneration minimally invasive surgery (Active Comparator): Periodontal regeneration minimally invasive surgery - Control Group 1
  Interventions: Procedure: Periodontal regeneration minimally invasive surgery
- Guided tissue regeneration surgery (Active Comparator): Guided tissue regeneration - Control Group 2
  Interventions: Procedure: Guided tissue regeneration surgery

INTERVENTIONS:
Device: Videoscope-assisted periodontal regeneration minimally invasive surgery — Use of a videoscope to improve visualization of periodontal defect during minimally invasive surgery
  Arms: Videoscope-assisted periodontal regeneration minimally invasive surgery
Procedure: Periodontal regeneration minimally invasive surgery — Conventional periodontal regeneration minimally invasive surgery without use of a videoscope
  Arms: Periodontal regeneration minimally invasive surgery
Procedure: Guided tissue regeneration surgery — Conventional guided tissue regeneration surgery for periodontal regeneration without use of a videoscope
  Arms: Guided tissue regeneration surgery

SUMMARY:
Clinical and preclinical studies confirm that regeneration of supporting tissues of teeth lost due to periodontal disease can be achieved using the principles of minimally invasive surgery (MIS). Although this therapeutic approach is well established in clinical settings and can rescue teeth with poor or questionable prognosis, MIS approaches often suffer from lack of predictability due to poor intraoral visibility of the bony lesion and inability to confirm thorough removal of etiological factors (plaque/calculus) on tooth surfaces. We seek to investigate whether improved visualization of the surgical field using an FDA approved videoscope (V) improves clinical outcomes. For this pilot study, N=50 (to attain 10/group) age, sex matched, systemically healthy subjects diagnosed with Stage III, Grade B periodontitis, formerly known as severe chronic periodontitis, will be randomly assigned to either the VMIS (Test), MIS (Control 1) or Guided Tissue Regeneration (GTR, Control 2) group. All periodontal therapy will be performed following the Standard of Care for periodontal regeneration to determine if utilization of the videoscope improves clinical and radiographic outcomes. We will examine bone fill using conventional digital periapical radiographs (PAR) and Cone Beam Computed Tomography (CBCT) imaging at 6 and 12 months compared to baseline and collect gingival crevicular fluid (GCF) to compare expression of growth factors and cytokines/chemokines during the healing period. This is a single center treatment study where subjects will be recruited from individuals seeking periodontal treatment at the Graduate Periodontics Clinic, UIC College of Dentistry (COD). Participation of all subjects will end after 12 months and will comprise 7 total visits.

ELIGIBILITY:
Inclusion Criteria:

* • Individual must be between the age of 18 and 70 years of age

  * ASA I or II systemically healthy subjects
  * Individuals presenting with at least 1 single or multirooted tooth with residual, isolated, interproximal bony defect with probing depths (PD) ≥ 6 mm, clinical attachment loss (CAL) ≥ 6mm, bleeding upon probing (BOP), and ≥ 2mm width of attached gingiva (WAG)
  * Radiographic evidence of interproximal alveolar bone loss, on existing (< 2 years old) dental radiographs of diagnostic quality taken at the COD
  * Vital tooth or previous root canal therapy with no signs/symptoms of pathology
  * Individuals with plaque scores ≤ 20%
  * English speaking subjects (Individual must be willing to follow all the study requirements and participate in the study procedures in its entirety and read, understand the informed consent form)

Exclusion Criteria:

* Individuals not referred from the Predoctoral Periodontics Student Clinics

  * Uncontrolled systemic disorders such as hypertension, heart disease, bleeding disorders, metabolic bone diseases, autoimmune disorders, etc., that may influence cellular/healing status
  * Diabetics
  * Current smokers
  * Individual less than 18 years of age
  * Individuals with non-isolated, interproximal PD ≥ 4 mm extending to the facial/buccal and/or palatal/lingual tooth surfaces
  * Teeth with Grade 2 or 3 mobility
  * Teeth with metal restorations such as a porcelain fused to metal crown (due to scattering of radiographic images)
  * Intrabony defects on dental implants
  * Individual who take medications known to affect host immunity or periodontal tissues (ex. steroids, antibiotics, phenytoin, etc.) in the previous 6 months
  * Individuals on chronic anti-platelet/anti-coagulant therapy
  * Oral pathologies other than periodontal disease (ex. periapical lesions of non-periodontal origin)
  * Subjects who may be pregnant based on a positive pregnancy test
  * Non-English speaking individuals

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | 6 months
  Measured in mm as the periodontal probing depth (PD) plus gingival recession (GR).
Probing Depth (PD) | 6 months
  Measured in mm as the distance from the gingival margin (GM) to the base of the gingival sulcus.
Gingival Recession (GR) | 6 months
  Measured in mm as distance of the gingival margin (GM) to the cemento-enamel junction (CEJ).
Radiographic Bone Height (RBH) | 6 months
  Measured in mm as the distance from the cemento-enamel junction (CEJ) to the base of the alveolar bone defect (ABD).
Radiographic Bone Volume (RBV) | 6 months
  Measured in cubic mm as the volume of bone from the alveolar crest (AC) to the base of the alveolar bone defect (ABD).
Clinical Attachment Level | 12 months
  Measured in mm as the periodontal probing depth (PD) plus gingival recession (GR).
Probing Depth (PD) | 12 months
  Measured in mm as the distance from the gingival margin (GM) to the base of the gingival sulcus.
Gingival Recession (GR) | 12 months
  Measured in mm as distance of the gingival margin (GM) to the cemento-enamel junction (CEJ).
Radiographic Bone Height (RBH) | 12 months
  Measured in mm as the distance from the cemento-enamel junction (CEJ) to the base of the alveolar bone defect (ABD).
Radiographic Bone Volume (RBV) | 12 months
  Measured in cubic mm as the volume of bone from the alveolar crest (AC) to the base of the alveolar bone defect (ABD).

SECONDARY OUTCOMES:
Gingival Crevicular Fluid (GCF) Growth Factor and Cytokine/Chemokine Levels | 6 months
  Concentration of 24 cytokines, chemokines, and growth factors in gingival crevicular fluid (GCF) measured in pg/mL.
Gingival Crevicular Fluid (GCF) Growth Factor and Cytokine/Chemokine Levels | 12 months
  Concentration of 24 cytokines, chemokines, and growth factors in gingival crevicular fluid (GCF) measured in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Nares, DDS, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, College of Dentistry, Periodontics, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No